CLINICAL TRIAL: NCT05150717
Title: Absorption, Distribution, Metabolism, and Excretion Study of [14C]-Jaktinib in Chinese Male Healthy Subjects(The Mass Balance and Biotransformation Study of [14C]-Jaktinib).
Brief Title: ADME Study of [14C]-Jaktinib in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK023
Record Dates: First submitted 2021-11-24; First posted 2021-12-09 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Healthy Adult Male Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-Jaktinib (Experimental): Subjects will receive single dose of [14C]-Jaktinib (Suspension, 100mg/150μCi)
  Interventions: Drug: [14C]-Jaktinib

INTERVENTIONS:
Drug: [14C]-Jaktinib — Subjects will receive single dose of orally [14C]-Jaktinib on Day 1.

SUMMARY:
This study was designed to evaluate the mass balance and biotransformation after single-dose of [14C]-Jaktinib orally in Chinese healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese males, aged 18-45 years old (inclusive);
* Body weight ≥ 50.0 kg, body mass index (BMI) between 19-26kg/m2 (inclusive);
* Sign the informed consent form；
* Participants are able to communicate well with the investigators and be able to complete the trial according to the Process.

Exclusion Criteria:

* Physical examination, vital signs, routine laboratory tests, 12-lead ECG, Chest X-ray, abdominal B-ultrasound and other is abnormal and clinically significant;
* Positive for hepatitis B surface antigen or E antigen, hepatitis C antibody, HIV antibody, or Treponema pallidum antibodies;
* Use of any prescription or over-the-counter drug, any vitamin product, health care drug or Chinese herbal medicine within 14 days prior to screening.
* Participants who have participated in any clinical trials within 3 months prior to screening and have used the test drug or medical devices.
* A history of any clinically serious illness or condition, including but not limited to circulatory, endocrine, nervous,digestive, urinary, or blood, immune, mental, and metabolic diseases, that the investigator considers to be likely to affect the results of the study.
* Participants who had heart disease such as heart failure, angina pectoris, myocardial infarction, and clinically significant arrhythmia.
* Participants who had undergone major surgery or whose surgical incision was not completely healed within 6 months before the screening period; Major surgery includes, but is not limited to, any surgery with a significant risk of bleeding, prolonged general anesthesia, or an open biopsy or significant traumatic injury.
* Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before screening.
* Hemorrhoids or perianal diseases with regular/bleeding in the stool; Patients with gastrointestinal dysfunction, such as irritable bowel syndrome and inflammatory bowel disease, may be affected by drug absorption as determined by researchers.
* Habitual constipation or diarrhea.
* Heavy drinking or regular drinking in the six months preceding the screening period, or alcohol breath test results ≥20 mg/dL during the screening period.
* Participants who had smoked more than 5 cigarettes per day on average in the 3 months before the screening period or habitually used nicotine-containing products and were unable to quit during the test period.
* Substance abuse or use of soft drugs (e.g., marijuana) in the 3 months prior to the screening period or use of hard drugs (e.g., cocaine, amphetamines, phenylcyclohexidine, etc.) in the 1 year prior to the screening period, or screening for positive urine drug abuse (drug) tests.
* Habitual consumption of grapefruit juice or excessive consumption of tea, coffee and/or caffeinated beverages and failure to abstain during the study period.
* Participants with a history of fainting needle or blood, have difficulty in blood collection or cannot tolerate vein puncture for blood collection.
* Workers engaged in conditions requiring long-term exposure to radioactivity; or have significant radiation exposure (≥2 chest/abdomen CT, or ≥3 other types of X-ray examinations) within 1 year before the test or have participated inthe radiopharmaceutical labeling test.
* Having family planning during the trial period and within 1 year after the last use of the drug, or not agreeing that subjects and their spouses should take strict contraceptive measures during the trial period and within 1 year after the last use of the drug.
* Participants who had lost blood or donated up to 400mL within 3 months before the screening period, or Participants who had received blood transfusion, or Participants who plan to donate blood within 3 month after the end of this test.
* As determined by the investigator, the subject has other factors that are not suitable for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion of 14C-labeled drug-related material (radioactivity in urine and fecal samples) | From the start of administration to 240 hours after administration
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in urine and feces.
Identification of the Proportion of different metabolites to determine biotransformation pathway of Jaktinib | From the start of administration to 240 hours after administration
  Proportion of different metabolites(Jaktinib and main metabolites)

SECONDARY OUTCOMES:
Quantitive analysis of the concentrations of Jaktinib and main metabolites in plasma to obtain pharmacokinetic data | From the start of administration to 240 hours after administration
  The concentrations of Jaktinib and main metabolites in plasma
Adverse events | From the start of administration to 17days after administration
  Adverse events assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: liyan Miao, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of soochow University, Suzhou, Jiangsu, China